CLINICAL TRIAL: NCT06642740
Title: Study on the Efficacy and Safety of Avatricopal in Patients With Chronic Liver Disease With Selective Invasive and Minimally Invasive Surgery Combined With Thrombocytopenia
Brief Title: Study on the Efficacy and Safety of Avatricopal in Patients With CLD Complicated With Thrombocytopenia
Status: Enrolling by invitation | Type: Observational
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, Head of Department, Beijing Ditan Hospital
Other Study IDs: DTXY29
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Liver Disease; Thrombopenia
MeSH Terms: conditions — Thrombocytopenia | interventions — Platelet Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Platelet count: <40×10^9/L: Subjects with platelet count <40×10^9/L will be given 60mg/ day of avatracopal
  Interventions: Other: Platelet count
- Platelet count :40-50×10^9/L: Subjects with platelet counts of 40-50×10^9/L will be given avatracopal 40mg/ day
  Interventions: Other: Platelet count

INTERVENTIONS:
Other: Platelet count — divide into two groups based on platelet count

SUMMARY:
In this study, patients with chronic liver disease undergoing selective invasive and minimally invasive surgery combined with thrombocytopenia were enrolled. After enrollment, liver disease treatment was supplemented with avatripopal for 5 days. Biochemical indexes of avatripopal were monitored during treatment and after withdrawal. The proportion of patients with platelet count ≥50×10^9/L on the day of selective invasive and minimally invasive surgery was analyzed. The incidence of adverse events was observed.

DETAILED DESCRIPTION:
This is a single-center, single-arm, prospective study. Patients with chronic liver disease undergoing selective invasive and minimally invasive surgery combined with thrombocytopenia. After enrollment, liver disease treatment was supplemented with avatripopal for 5 days. The baseline demographic data and biochemical data of the subjects were collected. Biochemical indexes of avatripopal were monitored during treatment and after withdrawal. The proportion of patients with platelet count ≥50×10^9/L on the day of selective invasive and minimally invasive surgery was analyzed. The incidence of adverse events was observed. To investigate the efficacy and safety of avatripopal in chronic liver disease patients with thrombocytopenia undergoing elective invasive and minimally invasive surgery. To provide reference for related clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily join the study and sign the informed consent;
* Age ≥18 years old, male or female;
* Baseline platelet count < 50×10^9/L;
* Patients with chronic liver disease undergoing elective invasive and minimally invasive surgery;
* No fertility requirements.

Exclusion Criteria:

* History of arterial or venous thrombosis within 6 months prior to baseline;
* Plan to receive platelet transfusion or platelet-containing blood products within 7 days prior to baseline visit;
* Anticoagulant or antiplatelet therapy cannot be suspended before surgery according to the standard (low-dose aspirin is allowed to continue);
* currently receiving treatment with recombinant human thrombopoietin or thrombopoietin receptor agonists (such as rhTPO, Etopopal, or romipristine);
* The subjects had severe arteriosclerosis, cerebral thrombosis tendency, coronary artery stenosis > 70%;
* Patients with a history of arterial or venous thrombosis within 6 months before enrollment;
* Patients with known portal vein blood flow velocity < 10 cm/s or previous portal vein thrombosis within 6 months before enrollment;
* Prior to enrollment, any known primary blood history (e.g., immune thrombocytopenia, myelodysplastic syndrome, aplastic anemia);
* A known history of hereditary prethrombotic syndrome prior to admission (e.g., VLeiden mutation, prothrombin G20210A mutation, or hereditary antithrombin III (ATIII) deficiency);
* A history of major cardiovascular disease within the 6 months prior to enrollment (e.g., aggravated congestive heart failure, arrhythmias known to increase the risk of thromboembolic events [such as atrial fibrillation], coronary or peripheral arterial stenting or angioplasty, and coronary or peripheral arterial bypass grafting);
* the subject is allergic to avatripopal or any of its excipients;
* Exclude vulnerable people with mental disorders and other disabilities
* The investigator believes that accompanying medical history may affect the safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease complicated with thrombocytopenia undergoing elective invasive and minimally invasive surgery were admitted to the experimental group for clinical observation.
Sampling Method: Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with platelet count ≥50×10^9/L on the day of elective invasive and minimally invasive surgery. | 2024-2025
  Proportion of patients with platelet count ≥50×10^9/L on the day of elective invasive and minimally invasive surgery.

SECONDARY OUTCOMES:
Adverse event rate | 2024-2025
  Recent and long-term thrombotic events and bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Yao Xie, Doctor, Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality, China